CLINICAL TRIAL: NCT03154229
Title: The Evaluation of a mHealth Platform for Diarrheal Disease Decision-support in Hospitals: a Cluster Randomized Controlled Trial
Brief Title: Evaluation of a mHealth Platform for Diarrheal Disease Decision-support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201601762 - N; 1DP5OD019893 (NIH); TW010182 [Pending] (Other Grant/Funding Number: John E. Fogarty International Center)
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Diarrhea
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paper-based decision-support (Active Comparator): Prior to starting the study, 10 hospitals will be made into 5 pairs. The paper versus smartphone intervention will be randomized to one member of each pair. The study arm will consist of a pre-interventional (6 weeks) followed by an interventional period (12 weeks); this arms will use paper-based decision support at the 5 hospitals designated.
  Interventions: Other: Paper-based decision-support; Other: Pre-Assessment of practices
- Smartphone-based decision-support (Active Comparator): Prior to starting the study, 10 hospitals will be made into 5 pairs. The paper versus smartphone intervention will be randomized to one member of each pair. The study arm will consist of a pre-interventional (6 weeks) followed by an interventional period (12 weeks); this arms will use smartphon-based decision support at the 5 hospitals designated.
  Interventions: Other: Smartphone-based decision-support; Other: Pre-Assessment of practices

INTERVENTIONS:
Other: Smartphone-based decision-support — WHO guidelines have been adapted from paper onto a smartphone referred to as a Rehydration Calculator
  Arms: Smartphone-based decision-support
Other: Paper-based decision-support — WHO guidelines presented on paper
  Arms: Paper-based decision-support
Other: Pre-Assessment of practices — Observation of baseline clinical practice.

SUMMARY:
The study hypothesis is that clinical decision-support on a smartphone for the management of diarrheal disease will improve the assessment of dehydration, reduce IV fluid usage, and increase guideline adherence for the use of zinc and antibiotics. To test this hypothesis we will conduct a cluster randomized controlled trial in the diarrhea wards of 10 hospitals in Bangladesh. A 6-week pre-intervention period will establish a baseline at all sites, and in the intervention, hospitals will be randomized to use a paper versus smartphone adaptation of the WHO guidelines by the admitting physician. Inclusion criteria are patients 2 months and older that have uncomplicated acute diarrheal disease; estimated enrollment is 7893 patients. The primary outcome measure is use of IV fluids. This project may have broad impact that will include opportunities to provide improved decision-support for the assessment of dehydration, decreased use intravenous fluids and more prudent use of antibiotics.

DETAILED DESCRIPTION:
Technology is making possible new approaches to overcome old public health challenges. Cellular networks are now ubiquitous in resource-poor settings and offer new opportunities for high-yield interventions for both chronic and acute diseases. We are specifically interested in developing mHealth solutions for diarrheal disease for two reasons. The first reason is that diarrheal disease globally remains the second leading cause of death for children less than 5 years of age. Barriers to combat this problem include poor adherence to guidelines for rehydrating children and outbreaks often outpace current epidemiological tools. The second reason is that diarrheal diseases in a setting like Bangladesh, including cholera outbreaks, are a model system to develop and test mHealth solutions that can be adapted to more complex chronic and acute diseases in Bangladesh and globally.

In partnership with the International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b; primary collaborator) and the Institute of Epidemiology, Disease Control, Research (IEDCR) within the Ministry of Health and Family Welfare in Bangladesh, we propose to compare a paper-based versus a smartphone-based decision-support tool in a cluster randomized controlled trial (cRCT) to determine the impact of the method of decision-support on the use of IV fluids (primary outcome) and indicated medications (secondary outcomes). The smartphone tool is an adaptation of the paper-based World Health Organization guidelines, and is called the 'Rehydration Calculator.' The cRCT will be conducted collaboratively between the icddr,b and government hospitals (N=10) in Bangladesh over 4.5 months per site. A 6-week pre-intervention period will establish a baseline at all sites, and in the intervention, hospitals will be randomized to use the paper versus smartphone tool by the admitting physician. Inclusion criteria are patients 2 months and older that have uncomplicated acute diarrheal disease; estimated enrollment is 7893 patients. Standard of care will be practiced at all sites, with the exception of the decision-support tool(s) in the interventional period. The primary outcome measure is use of IV fluids. This project may have broad impact that will include opportunities to provide improved decision-support for the assessment of dehydration, decrease intravenous fluid use and improve antibiotic stewardship.

ELIGIBILITY:
Inclusion Criteria:

* Acute uncomplicated diarrhea (less than 7 days with at least 3 loose stools in the last 24 hours)
* Age greater than or equal to two months.

Exclusion Criteria:

* No diarrhea
* Complicated diarrheal disease (e.g. e.g. sepsis, meningitis, convulsions, electrolyte imbalance, myocardial infarction, respiratory failure, chronic kidney disease, severe malnutrition by clinical measures and mid-upper arm circumference (<11.5cm for >= 6 mo to less than 5 years; <11.0 cm for >= 2mo to <6 mo))

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4975 (Actual)
Dates: Start 2018-03-11 (Actual); Primary Completion 2018-09-23 (Actual); Study Completion 2018-09-23 (Actual)

PRIMARY OUTCOMES:
Use of IV fluid | Intervention is 3 months per hospital
  The percentage of patients prescribed IV fluid between the paper-based decision-support and the Smartphone decision-support.

SECONDARY OUTCOMES:
Use of zinc | Intervention is 3 months per hospital
  The percentage of patients under five years prescribed zinc between the paper-based decision-support and the Smartphone decision-support.
Use of indicated antibiotics | Intervention is 3 months per hospital
  The percentage of patients prescribed the indicated antibiotic over 2 years of age that have acute watery diarrhea and severe dehydration between the paper-based decision-support and the Smartphone decision-support.

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Nelson, MD PhD, Principal Investigator — University of Florida, USA
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh (icddr,b), Dhaka, Dhaka Division, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haque F, Ball RL, Khatun S, Ahmed M, Kache S, Chisti MJ, Sarker SA, Maples SD, Pieri D, Vardhan Korrapati T, Sarnquist C, Federspiel N, Rahman MW, Andrews JR, Rahman M, Nelson EJ. Evaluation of a Smartphone Decision-Support Tool for Diarrheal Disease Management in a Resource-Limited Setting. PLoS Negl Trop Dis. 2017 Jan 19;11(1):e0005290. doi: 10.1371/journal.pntd.0005290. eCollection 2017 Jan. PMID 28103233
- [Derived] Khan AI, Mack JA, Salimuzzaman M, Zion MI, Sujon H, Ball RL, Maples S, Rashid MM, Chisti MJ, Sarker SA, Biswas D, Hossin R, Bardosh KL, Begum YA, Ahmed A, Pieri D, Haque F, Rahman M, Levine AC, Qadri F, Flora MS, Gurka MJ, Nelson EJ. Electronic decision support and diarrhoeal disease guideline adherence (mHDM): a cluster randomised controlled trial. Lancet Digit Health. 2020 May;2(5):e250-e258. doi: 10.1016/S2589-7500(20)30062-5. PMID 33328057
- See also: Pilot study publication — http://journals.plos.org/plosntds/article?id=10.1371/journal.pntd.0005290